CLINICAL TRIAL: NCT01781104
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multiple Dose, Parallel Group Study to Evaluate the Efficacy, Safety, and Pharmacodynamics of RM-131 Administered to Patients With Chronic Constipation
Brief Title: Phase 2 Study to Evaluate Safety and Efficacy of RM-131 Administered to Patients With Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM-131-006
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Constipation
Keywords: constipation gastric emptying gastrointestinal motility ghrelin
MeSH Terms: conditions — Constipation | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RM-131 (Active Comparator)
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131 — Double blind RM-131 (100 ug) will be delivered subcutaneously once daily for 14 days.
  Arms: RM-131
Drug: Placebo — Placebo delivered subcutaneously once daily for 14 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability as well as the effects of RM-131 on colonic transit, bowel consistency, bowel habits, abdominal pain, and other abdominal symptoms in patients with chronic constipation.

ELIGIBILITY:
Inclusion criteria

* Able to provide written informed consent prior to any study procedures, and willing and able to comply with study procedures.
* Diagnosis of chronic IDIOPATHIC constipation, including experiencing constipation for 12 or more weeks in the preceding 12 months (defined by Rome III criteria for Functional Constipation, but all patients must meet the modified criterion of a history of ≤4 average defecations per week)
* Stable concomitant medications (no changes in regimen for at least 2 weeks prior to baseline period)
* Body mass index of 18-40 kg/m2
* Females must not be lactating or pregnant

Exclusion criteria

* Unable/unwilling to provide informed consent or to comply with study procedures
* Diagnosis of secondary constipation e.g. underlying general neurological disease such as Parkinsonism, multiple sclerosis, diseases associated with peripheral neuropathy, iatrogenic constipation
* Structural or metabolic diseases that affect the GI system NOTE: Patients with clinical suspicion of upper or lower GI obstruction must have been evaluated per standard of care and obstruction ruled out before screening
* Unable to withdraw the following medications 48 hours prior to baseline period and throughout the study (except as protocol defined rescue medications):

  * Medications that alter GI transit including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin, narcotics, anti-cholinergics, tricyclic antidepressants, SNRI and newer antidepressants
  * Selective serotonin reuptake inhibitor (SSRI) antidepressants are permissible at low, stable doses
  * Analgesic drugs including opiates, NSAIDs and COX-2 inhibitors
  * GABAnergic agents
  * Benzodiazepines
* NOTE: stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection, and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible
* Drugs with a low therapeutic index, such as warfarin, digoxin, anti-seizure medications
* History of surgery within 60 days of screening
* Acute or chronic illness or history of illness, which in the opinion of Investigator, could pose threat/harm to the patient or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc
* History of hypersensitivity to mannitol (an ingredient of both active and placebo study medications)
* Clinically significant abnormalities on screening laboratories or physical examination as determined by Investigator
* Abnormal 12-lead electrocardiogram (ECG), including evidence of acute myocardial or subendocardial ischemia and clinically significant arrhythmias or conduction abnormalities (including prolonged QTc > 500 msec) or abnormal blood pressure at screening except minor deviations deemed to be of no clinical significance by Investigator
* Acute GI illness within 48 hours of initiation of the baseline period
* ALT or AST > 1.2 X upper limit of normal during screening
* Females who are pregnant or breastfeeding
* History of excessive alcohol use or substance abuse
* Participation in an investigational clinical study within 30 days prior to dosing in the present study
* Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study

Exclusion criteria at the end of the baseline period

* In addition, patients will not be randomized into the double-blind treatment comparison if during the baseline period they:
* used rescue medications such as laxatives, beyond those allowed by protocol
* demonstrated lack of compliance
* averaged more than 4 spontaneous bowel movements per week
* Substudy patients only: did not demonstrate slow colonic transit at end of baseline period (GC 24 >2.4)
* Women of child-bearing potential: positive pregnancy test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Effect of RM-131 on colonic transit | End of 14 day Baseline and end of 14 day Treatment periods
  Change from baseline colonic geometric center at 24 hours

SECONDARY OUTCOMES:
Safety and tolerability of RM-131 | Duration of the study, an expected average of 9 weeks
  Assessment of adverse events and clinical laboratory evaluations
Effect of RM-131 on stool consistency | Daily for the duration of the study, an expected average of 9 weeks
  Change in responses on Bowel Habit Diary Cards

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stoner, MD, Study Director — Rhythm Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Acosta A, Camilleri M, Busciglio I, Boldingh A, Nelson AD, Burton D. Short-Term Effects of Relamorelin on Descending Colon Motility in Chronic Constipation: A Randomized, Controlled Trial. Dig Dis Sci. 2016 Mar;61(3):852-60. doi: 10.1007/s10620-015-3876-5. Epub 2015 Oct 14. PMID 26467700
- [Derived] Acosta A, Camilleri M, Kolar G, Iturrino J, Szarka LA, Boldingh A, Burton D, Ryks M, Rhoten D, Zinsmeister AR, Spence SC, Gottesdiener K, Bouras EP, Vazquez-Roque MI. Relamorelin Relieves Constipation and Accelerates Colonic Transit in a Phase 2, Placebo-Controlled, Randomized Trial. Clin Gastroenterol Hepatol. 2015 Dec;13(13):2312-9.e1. doi: 10.1016/j.cgh.2015.04.184. Epub 2015 May 19. PMID 26001337